CLINICAL TRIAL: NCT04620954
Title: A Phase I/II Clinical Trial to Evaluate Platinum-based Chemotherapy, Oregovomab and Nivolumab in Patients With Platinum Sensitive Recurrent Epithelial Cancer of Ovarian, Tubal or Peritoneal Origin
Brief Title: Clinical Trial of Chemotherapy, Oregovomab and Nivolumab in Patients With Epithelial Cancer of Ovarian, Tubal or Peritoneal Origin
Acronym: ORION-02
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: CanariaBio Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC OV-03
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2020-12

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — oregovomab; Nivolumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Drug: Oregovomab; Drug: Nivolumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Oregovomab — 2mg of Oregovomab is administered through IV on Weeks 1, 5, 9, 17.
Drug: Nivolumab — 480mg of Nivolumab is administered through IV every 4 weeks (Weeks 9, 13, 17, 21).
Drug: Chemotherapy — Pegylated liposomal doxorubicin (PLD) and carboplatin are administered every 4 weeks through IV. The starting dose of PLD and carboplatin are 30mg/m^2 and 5 AUC (Area Under the Curve) respectively.

SUMMARY:
This is an open-label, single-arm, phase I/II, single-center study with dose finding and dose expansion parts.

This study hypothesizes that the combination of platinum-based chemotherapy, Oregovomab and Nivolumab will improve intracellular CA 125 antigen processing and elicit a stronger systemic CA 125-specific T cell response and that it will be in a manner that is synergistic, safe and clinical efficacious in patients with relapsed platinum sensitive epithelial ovarian carcinoma (EOC).

ELIGIBILITY:
Inclusion Criteria:

Signed Written Informed Consent

* Able to understand and voluntarily sign the Informed Consent Form (ICF). Written informed consent must be obtained before any study specific procedures that are not part of standard of care.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory test, and other protocol requirements
* Age ≥ 21 years old

Age and Target Population

* Histologically and/or cytologically confirmed diagnosis of epithelial ovarian, fallopian tube and primary peritoneal carcinoma (including carcinosarcoma)
* Serum CA 125 level at enrollment must be at least 5 times the upper limit of normal (ULN) using local laboratory ranges
* Objective evidence of disease progression after 2 to 3 prior lines of cytotoxic chemotherapy including (neo)adjuvant platinum-based regimen for advanced stage disease. Patients may have received prior treatment with Bevacizumab and/or poly ADP ribose polymerase (PARP) inhibitor in any line, including as maintenance therapy.
* Disease progression occurring at least 6 months after the last dose of platinum therapy was given following the penultimate line of chemotherapy before enrollment
* Presence of:

  1. measurable disease as defined by RECIST v1.1 AND a pre-treatment serum CA 125 level ≥ 5 times ULN on 1 occasion, OR
  2. non-measurable but evaluable disease such as ascites and pleural effusions attributable to disease or radiologic abnormalities that do not meet RECIST v1.1 criteria AND a pre-treatment serum CA 125 level ≥ 5 times ULN on 2 occasions at least 1 week apart, OR
  3. non-evaluable, non-measurable disease as defined by RECIST v1.1 AND pre- treatment CA 125 level ≥ 5 times ULN on 2 occasions at least 1 week apart
* Estimated life expectancy greater than 3 months
* Performance status Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Adequate hematologic and end organ function, defined by the following local laboratory results obtained within 14 days before study entry:

  1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks of laboratory test used to determine eligibility)
  2. White Blood Cell (WBC) count ≥ 2.0 × 109/L
  3. Platelet count ≥ 100 × 109/L (without transfusion within 2 weeks of laboratory test used to determine eligibility)
  4. Hemoglobin ≥ 9.0 g/dL
  5. Creatinine clearance (CrCl) ≥ 30 ml/min according to Cockcroft-Gault formula
  6. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 3 x ULN (or ≤ 5 x ULN in patients with liver metastases)
  7. Serum bilirubin ≤ 1.5 x ULN (except patients with known Gilbert's disease who have serum bilirubin level ≤ 3 x ULN)
* Normal Thyroid Stimulating Hormone (TSH) and free Thyroxine (fT4) levels
* Recovery of acute AEs of prior anticancer therapies, including surgery and radiotherapy, to baseline or CTCAE grade ≤ 1 before study entry

Reproductive Status

* Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of hCG) within 24 hours before study entry
* No breastfeeding
* WOCBP must agree to observe abstinence from heterosexual sexual intercourse, or use contraceptive methods that results in a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of Nivolumab.

Exclusion Criteria:

Cancer-specific Exclusions

* Non-epithelial ovarian tumors or ovarian tumors with low malignant potential (i.e., borderline tumors). Note: ovarian carcinosarcomas are eligible.
* Active symptomatic central nervous system (CNS) metastases. Patients with previous CNS metastases are eligible provided that they underwent CNS irradiation, are asymptomatic, do not require treatment with radiation therapy or anticonvulsants, and have stable disease at the screening tumor assessment. In addition, these patients must have been either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisolone (or equivalent).
* Spinal cord compression not definitively treated with surgery and/or radiation. Patients with previously diagnosed and treated spinal cord compression are eligible provided that they have stable disease at the screening tumor assessment. In addition, these patients must have been either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisolone (or equivalent).
* Leptomeningeal carcinomatosis
* Uncontrolled pleural effusion(s), pericardial effusion or ascites requiring recurrent drainage procedures (Patients with functioning pleural and/or peritoneal drainage catheters/devices in situ at time of study entry may be eligible.)
* Previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 2 years before study entry AND no additional therapy is required, or anticipated to be required, during the study period

General Medical Exclusions

* Pregnant or lactating women
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months before study entry, unstable arrhythmias/heart block, or unstable angina
* Severe infections within 4 weeks before study entry including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* History of abdominal fistula, history of gastrointestinal perforation, and signs or symptoms of bowel obstruction
* Symptoms or radiological evidence of active bowel obstruction
* Non-healing wound or ulcer, or bone fracture within 3 months before study entry.
* Concurrent anticancer treatment within 28 days before study entry, e.g. cytotoxic chemotherapy, radiotherapy (except for palliative bone-directed radiotherapy), immunotherapy, cytokine therapy (except for erythropoietin); major surgery within 28 days before study entry (excluding diagnostic biopsy); use of hormonal agents within 7 days before study entry; or use of any investigational drug within 28 days before study entry. Patients receiving bisphosphonate or denosumab are eligible provided treatment was initiated at least 14 days before study entry.
* Seizure disorder requiring anti-epileptic medication
* Renal failure requiring hemo- or peritoneal dialysis
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or administration of Investigational Products (IPs), or interfere with the interpretation of safety results
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Exclusions Related to Investigational Products

* Other concurrent/ongoing systemic investigational agents
* Previous assignment to treatment during this study. Subjects permanently withdrawn from study treatment participation will not be allowed to re-enter the study.
* History of severe allergic, anaphylactic or other hypersensitivity reactions attributed to murine or humanized antibodies or fusion protein, biopharmaceuticals produced in Chinese hamster ovary cell products, or compounds of similar chemical or biologic composition to platinum(s), PLD, Oregovomab or Nivolumab
* Prior treatment with anti-CA 125 cancer vaccine, or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA 4) antibody or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Active, known or suspected autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Subjects with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded.
* Active use of systemic corticosteroids (≥ 10mg/day prednisolone or equivalent) or other systemic immunosuppressive agents (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF) agents) within 7 days before study entry, or anticipated requirement for systemic immunosuppressive medications during the study, with the following exceptions:

  1. Systemic corticosteroids at physiologic doses to treat adrenocortical insufficiency not to exceed 10 mg/day of prednisolone or equivalent
  2. Steroids as premedication for hypersensitivity reactions (e.g. premedication for Carboplatin, PLD or CT contrast medium)
  3. Intranasal, inhaled, ophthalmic topical glucocorticoids, local (e.g. intra-articular) steroid injections, and systemic mineralocorticoids (e.g. fludrocortisone)
* History of solid organ allograft or allogeneic hematopoietic stem cell transplantation
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen (HBsAg) test and a positive antibody to hepatitis B core antigen (anti-HBc) antibody test) are eligible. Patients with hepatitis B (HBV) infection (defined as having a positive HBsAg test) AND undetectable HBV DNA titer are also eligible.
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks before study entry, or anticipation that such a live attenuated vaccine will be required during the study
* Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity

Other Exclusions Criteria

- Inability to attend or comply with treatment of follow-up scheduling

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Number of incidences of adverse events (AE) | From time of start of treatment to the date of disease progression or death due to any cause, up to 2 years
Proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) | From time of start of treatment to CR or PR, up to 2 years
  Objective response rate

SECONDARY OUTCOMES:
Proportion of patients with best overall response of CR, PR, or Stable Disease (SD) | From time of start of treatment to CR, PR or SD, up to 2 years
  Disease control rate
Progression free survival | From time of start of treatment to first documented progression or death due to any cause, up to 2 years
Overall survival | From time of start of treatment to time of death due to any cause, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jack Chan, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Center Singapore, Singapore